CLINICAL TRIAL: NCT06069336
Title: Nebulised 3% Hypertonic Saline Versus 0.9% Saline for Treating Patients Hospitalized With Acute Bronchiolitis: Protocol of a Randomized, Double-blind, Multicentre Trial
Brief Title: Nebulised 3% Hypertonic Saline Versus 0.9% Saline for Treating Patients Hospitalized With Acute Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szpital im. Św. Jadwigi Śląskiej (Other)
Responsible Party: Principal Investigator, Henryk Szymański, Head of Paediatric Department, Szpital im. Św. Jadwigi Śląskiej
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1/2023
Record Dates: First submitted 2023-09-23; First posted 2023-10-05 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Bronchiolitis
Keywords: hypertonic saline; infants; RCT
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomization will occur within 24 hours of admission
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypertonic saline (Active Comparator): 3% hypertonic saline (NEBU-dose hypertonic). The treatment will be delivered through nebulisation using oxygen with 5 litres of O2 flow, or through a compressed air-driven jet nebuliser, every 6 hours for three times daily with a night break, until discharge.
  Interventions: Drug: Hypertonic saline
- Normal saline (Placebo Comparator): 0,9% normal saline (NEBU-dose isotonic).The treatment will be delivered through nebulisation using oxygen with 5 litres of O2 flow, or through a compressed air-driven jet nebuliser, every 6 hours for three times daily with a night break, until discharge.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Hypertonic saline — Nebulised 3% hypertonic saline (NEBU-dose hypertonic). Nebulisation will be performed by trained study nurses or by parents under the supervision of a nurse
  Arms: Hypertonic saline
Drug: Normal saline — 0,9% normal saline (NEBU-dose isotonic). Nebulisation will be performed by trained study nurses or by parents under the supervision of a nurse
  Arms: Normal saline

SUMMARY:
Bronchiolitis is an acute viral infection of the lower respiratory tract. It is most commonly caused by respiratory syncytial virus (RSV). Only supportive therapy, including suctioning nasal secretions, water-electrolyte balance maintenance, and oxygen supplementation when needed, is recommended. The inhalation of 3% hypertonic saline is not recommended in bronchiolitis management. However, a recently published meta-analysis revealed that the inhalation of hypertonic saline can reduce the risk of hospitalisation for outpatients with bronchiolitis, while resulting in a shorter length of hospital stay and reduced severity of respiratory distress for inpatients, although the evidence is of low certainty.

The aim of the study is to assess the efficacy of nebulised hypertonic saline for the treatment of children hospitalised with bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

1. Children admitted to the hospital with the clinical diagnosis of acute bronchiolitis, which is defined as an apparent viral respiratory tract infection associated with airway obstruction manifested by at least one of following symptoms:

   * Tachypnoea (WHO definition).
   * Increased respiratory effort manifested as follows:

     1. Nasal flaring;
     2. Grunting;
     3. Use of accessory muscles;
     4. Intercostal and/or subcostal chest wall retractions;
     5. Apnoe.
   * Crackles and/or wheezing.
2. Aged 5 weeks - 24 months old.
3. A caregiver must provide written informed consent.

Exclusion Criteria:

1. Infants hospitalised with severe bronchiolitis (requiring mechanical ventilation or intensive care, or oxygen saturation < 85% on room air).
2. History of prematurity (gestational age <34 weeks).
3. Diagnosis of a clinically significant chronic disease (cardiac, respiratory, neuromuscular, or metabolic).
4. Immunodeficiency.
5. Gastro-oesophageal reflux.
6. Diagnosis or suspicion of asthma.
7. Inhaling a nebulised 3% hypertonic saline solution within 12 hours before enrolment.
8. Inhaling bronchodilators within 24 hours before enrolment.
9. Inhaling steroids within 24 hours before enrolment.
10. Systemic steroid therapy in the preceding 2 weeks.

Ages: 5 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay (LOS). | From admission to hospital discharge

SECONDARY OUTCOMES:
Number of participants requiring oxygen supplementation | During the intervention
Duration of oxygen supplementation | During the intervention
  among those requiring oxygen
The time until the infant will be assessed as being 'fit for discharge' | During the intervention
  which is defined as the point at which the infant will be feeding adequately (taking >75% of their usual intake based on parents' assessment) and will have a saturation of at least 92% for 6 h on room air, while the axillary body temperature will remain - among those requiring oxygen
Number of participants requiring hospital readmission after discharge | 7 days after the end of interventions
Number of adverse events | 7 days after the end of interventions
  especially incidence of acute otitis media and pneumonia
Worsening of clinical status, including the following: | During the intervention
  PICU admission The need for oxygen supplementation via HNFC; Bronchospasm within 30 minutes of a nebulised study treatment as indicated by an increase/worsening of the RDAI of <4 points.
Value of clinical severity score (RDAI and Wang Scale) | During the intervention
  30 minutes after intervention and 24 h, 48 h, and 72 h after enrolment

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - Szpiatal im.Świętej Jadwigi Śląskiej, Trzebnica
  - Dziecięcy Szpital Kliniczny im. Polikarpa Brudzińskiego w Warszawie, Warsaw
  - Specjalistyczny Szpital im. Alfreda Sokołowskiego w Wałbrzychu, Wałbrzych

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or generated during this study will be made available after the publication of results
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Avaliable after the publication
Access Criteria: Upon researcher's personal request

REFERENCES:
- [Derived] Szupienko S, Buczek A, Szymanski H. Nebulised 3% hypertonic saline versus 0.9% saline for treating patients hospitalised with acute bronchiolitis: protocol for a randomised, double-blind, multicentre trial. BMJ Open. 2023 Nov 27;13(11):e080182. doi: 10.1136/bmjopen-2023-080182. PMID 38011984